CLINICAL TRIAL: NCT03475654
Title: Virtual-Environment Home Rehabilitation: a Randomized Controlled Trial
Brief Title: A Prospective Trial of Virtual Home Rehabilitation After Burn Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Tam Pham, Professor, School of Medicine: Surgery: Trauma, Burn and Critical Care Division, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00003707
Record Dates: First submitted 2018-03-01; First posted 2018-03-23 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Burns; Burn Scar; Contracture
Keywords: exercise; therapy; rehabilitation; home
MeSH Terms: conditions — Burns; Contracture; Motor Activity

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- technology-assisted rehabilitation (Experimental): The experimental group will receive treatment as usual, in addition to training with the Jintronix platform. Participants will undergo their prescribed therapy regimen for 3 months, with outcomes follow-up to 12 months post-discharge.
  Interventions: Behavioral: Technology-assisted rehabilitation
- Usual care (Active Comparator): The control group will receive treatment as usual, which includes a personalized home exercise program prescribed by a burn therapist, prior to hospital discharge. Participants will undergo their prescribed therapy regimen for 3 months, with outcomes follow-up to 12 months post-discharge.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Technology-assisted rehabilitation — The Jintronix software platform, coupled with the Microsoft Kinect for movement capture, contains individualized exercise modules to increase ROM, endurance and strength. Within this PRCT, online monitoring of activity and actigraphy measurements through a wearable device and completion of an online diary will provide enhanced monitoring of home activities.
  Arms: technology-assisted rehabilitation
Behavioral: Usual care — The control group will receive treatment as usual, which includes a personalized home exercise program prescribed by a burn therapist, prior to hospital discharge.
  Arms: Usual care

SUMMARY:
The overarching goal for this prospective randomized controlled trial (PRCT) is to determine whether a virtual-environment, home-rehabilitation program improves functional outcomes for individuals after a burn injury. Specifically, this study will test the efficacy of a technology-assisted rehabilitation program against current standard of home therapy.

DETAILED DESCRIPTION:
This is a prospective, randomized controlled trial (PRCT) involving 50 adult burn survivors. This study tests the efficacy of a technology-assisted rehabilitation program against current standard of home therapy. There are two study groups for which subjects will be randomized: control and experimental.The control group will receive treatment as usual, which includes a personalized home exercise program prescribed by a burn therapist, prior to hospital discharge. The experimental group receives treatment as usual, in addition to training and use of the Jintronix platform for 3 months after hospital discharge. Participants will undergo their prescribed therapy regimen for 3 months, with outcomes follow-up to 12 months post-discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years old (no upper age limit)
* Ability to provide written, informed consent for study participation
* Ability to read and understand English
* Anticipated discharge to home environment
* Home environment includes access to:

  * television (larger than 20 inches in diameter with High Definition Multimedia Interface input (HDMI)
  * internet and email address
  * telephone (cell phone or landline)

Exclusion Criteria:

* Age less than 18 years
* Inability to provide written, informed consent for study participation
* Inability to read or understand English
* Delirium (as determined by the Delirium Observation Score test)
* Near-fall event at time of screening
* Pregnant women
* Discharge to non-home environment (e.g., shelter, street, skilled nursing facility)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Level of physical activity | 3 months after study enrollment
  level of activity among enrolled subjects by actigraphy

SECONDARY OUTCOMES:
Range of motion (ROM) | Study enrollment, 3, 6 and 12 months after enrollment
  ROM by subjects in each group
Patient-reported outcome measures (PROMIS): sleep | Study enrollment, 3, 6, 12 months after enrollment
  Sleep and sleep disturbance Short Form (SF)8B PROMIS tool
Patient-reported outcome measures (PROMIS): social participation | Study enrollment, 3, 6, 12 months after enrollment
  Participation in social roles and activities PROMIS tool SF6A
Patient-reported outcome measures (PROMIS): pain interference | Study enrollment, 3, 6, 12 months after enrollment
  Pain interference PROMIS tool SF6A
Patient-reported outcome measures (PROMIS): fatigue | Study enrollment, 3, 6, 12 months after enrollment
  Fatigue PROMIS tool SF6A
Patient-reported outcome measures (PROMIS): stiffness | Study enrollment, 3, 6, 12 months after enrollment
  Stiffness impact Adult Sickle Cell Quality of Life Measurement Information System (ASCQ-ME) V2.0
Patient-reported outcome measures (PROMIS): mobility | Study enrollment, 3, 6, 12 months after enrollment
  Mobility PROMIS tool
Patient-reported outcome measures (PROMIS): upper extremity | Study enrollment, 3, 6, 12 months after enrollment
  Upper extremity PROMIS SF7A
Return to work/school | up to 1 year
  Date when subject returns to work or school
Patient reported level of activity difficulty | Weekly beginning 1 week after study enrollment and concluding 3 months after study enrollment
  Using 1-5 difficulty scale (1=no difficulty and 5=very difficult), subject is asked how difficult his/her activity has been for the past 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Tam Pham, MD, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No